CLINICAL TRIAL: NCT06411028
Title: Factors Determining the Efficacy of Botulinum Toxin for Arm Tremor in Dystonia: An Exploratory Study
Brief Title: Factors Determining the Efficacy of Botulinum Toxin for Arm Tremor in Dystonia
Acronym: BAT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); Donders Centre for Cognitive Neuroimaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115083; 2024-515970-28 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Dystonic Tremor Syndrome
Keywords: Botulinum neurotoxin; Botulinum toxin; Dystonia; Dystonic tremor syndrome; Dystonic tremor; Tremor associated with dystonia; Upper extremity; Functional magnetic resonance imaging; fMRI; Muscle ultrasound
MeSH Terms: conditions — Dystonia | interventions — Magnetic Resonance Imaging; Botulinum Toxins

STUDY DESIGN:
Intervention Model Description: Uncontrolled multi-centre low-intervention clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botulinum toxin (Experimental): Participants are treated with three consecutive BoNT sessions.
  Interventions: Diagnostic Test: Polymyography; Diagnostic Test: Muscle ultrasound; Diagnostic Test: (Functional) magnetic resonance imaging; Diagnostic Test: Clinical assessment; Diagnostic Test: Questionnaires; Drug: botulinum toxin injection (BTX A)

INTERVENTIONS:
Diagnostic Test: Polymyography — We will measure muscle activity using surface electromyography and tremor using inertial measurement units while subjects perform rest, posturing and kinetic tasks.
  Other Names: Tremor registration; Poly-electromyography
Diagnostic Test: Muscle ultrasound — We will obtain B-mode images and videos of upper extremity muscles of the most affected upper extremity.
Diagnostic Test: (Functional) magnetic resonance imaging — Subjects will undergo (f)MRI scanning involving concurrent electromyography, accelerometry and functional magnetic resonance imaging.
Diagnostic Test: Clinical assessment — We will assess tremor and dystonia severity using clinical scales.
Diagnostic Test: Questionnaires — We will collect patient-reported outcomes.
Drug: botulinum toxin injection (BTX A) — Three consequetive botulinum toxin injections of the upper extremities

SUMMARY:
Tremor occurs in up to 55% of dystonia patients, which is known as dystonic tremor syndrome (DTS). Tremor can be present in the body part affected by dystonia (dystonic tremor, DT), or an unaffected body part (tremor associated with dystonia, TAWD). DTS can be treated with botulinum neurotoxin (BoNT) injections, but BoNT is effective in only about 60-70% of patients. It is unknown which patients benefit most from BoNT treatment. The investigators aim to explore the associations between clinical and pathophysiological tremor characteristics and BoNT efficacy. To do so, the investigatorswill measure clinical, electrophysiological, ultrasonographic and (functional) magnetic resonance imaging ((f)MRI) characteristics before the start of BoNT treatment and measure BoNT efficacy after three three-monthly BoNT sessions.

DETAILED DESCRIPTION:
Rationale: Tremor occurs in up to 55% of dystonia patients, which is known as dystonic tremor syndrome (DTS). Tremor can be present in the body part affected by dystonia (dystonic tremor, DT), or an unaffected body part (tremor associated with dystonia, TAWD). DTS can be treated with botulinum neurotoxin (BoNT) injections, but BoNT is effective in only about 60-70% of patients. It is unknown which patients benefit from BoNT treatment. This highlights the need for personalized treatment.

Objective: The primary objective is to explore the associations between clinical, electrophysiological, ultrasonographic and (functional) magnetic resonance imaging ((f)MRI) tremor characteristics and BoNT efficacy in DTS of the upper extremity. The secondary objectives are to:

* Explore the clinical, electrophysiological, ultrasonographic and (f)MRI differences between DT and TAWD of the upper extremity.
* Explore the agreement between a clinical assessment, polymyography (PMG) and muscle ultrasound (MUS) on muscle selection in DTS of the upper extremity.

Study design: An uncontrolled multi-centre low-intervention clinical trial where subjects participate for ± 8 months Study population: 60 adults with DTS (± 30 DT/ 30 TAWD) of the upper extremity who start 12-weekly BoNT treatment in normal clinical practice.

Main study parameters/endpoints: the associations between clinical, electrophysiological, ultrasonographic, and (f)MRI tremor characteristics at baseline and BoNT efficacy (change in TRG Essential Tremor Rating Assessment Scale (TETRAS) from baseline to 28 weeks).

Secondary trial endpoints:

* The clinical, electrophysiological, ultrasonographic and (f)MRI differences between DT and TAWD at baseline.
* The agreement between a clinical assessment, PMG and MUS on muscle selection. Intervention: Participants are treated with three consecutive BoNT sessions in normal clinical practice. Participants will undergo additional diagnostic procedures: 2 clinical assessments, 2 PMGs, 1 MUS recordings and 1 fMRI assessment and will fill in 2 questionnaires before and after the BoNT sessions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of dystonic tremor or tremor associated with dystonia according to the 2018 consensus statement on the classification of tremors
* Tremor of one or both upper extremities
* Starting botulinum toxin injections as part of normal clinical practice
* Age ≥ 18 years

Exclusion Criteria:

* Acquired aetiology of dystonic tremor syndrome
* Previous botulinum toxin treatment of the to be treated upper extremity for ≥ 4 consecutive sessions
* In case of previous botulinum toxin treatment of the to be treated upper extremity for ≤3 consecutive sessions: the last botulinum toxin injections ≤ 6 months before study enrolment
* Unstable dose medications for dystonia and tremor ≤ 1 month before study enrolment
* Deep brain stimulation implantation ≤ 6 months before study enrolment
* Unstable deep brain stimulation variables ≤ 1 month before study enrolment
* Comorbidity interfering with study participation
* Known hypersensitivity for components of Dysport
* Infection at the upper extremity
* Pregnancy, trying to conceive and breastfeeding
* Insufficient knowledge of the Dutch or English language

Exclusion criteria for MRI scanning:

* Contraindications for MRI (e.g. previous brain surgery, claustrophobia, active implant, epilepsy, metal objects in the upper body that are incompatible with MRI)
* Moderate to severe head tremor while lying supine (to avoid artefacts caused by extensive head motion during scanning).
* Inability to provoke postural tremor while lying supine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Tremor severity assessed by the TRG Essential Tremor Rating Assessment Scale (TETRAS) | Baseline, 28 weeks
  The primary outcome is the clinical tremor severity measured by the TRG Essential Tremor Rating Assessment Scale (TETRAS) at 28 weeks. The scale ranges between 0 and 112 points, with higher scores indicating a more severe tremor. The TETRAS consists of two subcategories: a 12-item activities of daily living subscale and a 9-item performance scale. The daily living subscale is scored by interviewing the participant. The performance scale is rated by observing the participants while they are performing multiple tasks.

SECONDARY OUTCOMES:
Tremor severity assessed by the Fahn-Tolosa-Marin Tremor Rating Scale (FTM-TRS) | Baseline, 28 weeks
  FTM-TRS [0-152]: higher scores indicate a more severe tremor.
Dystonia severity assessed by the Burke-Fahn-Marsden Dystonia Rating Scale (BFM-DRS) | Baseline, 28 weeks
  BFM-DRS [0-150]: higher scores indicate more severe dystonia.
Additional neurological signs assessed by the Standardised Tremor Elements Assessment (STEA) | Baseline
  STEA [0-27]: higher scores make a diagnosis of dystonic tremor syndrome instead of essential tremor more likely.
Quality of life assessed by the Quality of Life Essential Tremor Questionnaire (QUEST) | Baseline, 28 weeks
  QUEST [0-120]: higher scores indicate greater dissatisfaction.
Psychological stress assessed by the Perceived stress scale (PSS) | Baseline, 28 weeks
  PSS [0-4]: higher scores indicate higher levels of perceived stress
Pain assessed by the Numeric Pain Rating Scale (NPRS) | Baseline, 28 weeks
  NPRS [0-10]: 0 indicates no pain and 10 the worst imaginable pain
Patient-reported change in tremor severity assessed by the Patient Global Impression of Change (PGIC) | 28 weeks
  PGIC [-3: much worse, -2: moderately worse, -1: slightly worse, 0: no change, 1: slightly better, 2: moderately better, 3: much better]
Electrophysiological characteristics | Baseline, 28 weeks
  e.g. tremor power, dominant frequency, frequency-width at half-width power, intermuscular coherence, tremulous muscles
Ultrasonographic tremulous activity | Baseline
Tremor related cerebral activity | Baseline
  Quantified using functional MRI scanning
Botulinum toxin parameters | Baseline, 12 and 24 weeks
  e.g. injection schemes, rationale for muscle selection, adherence

CONTACTS AND LOCATIONS:
Overall Officials: Anke Snijders, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Donders Centre for Cognitive Neuroimaging, Nijmegen, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymised participant data will be shared in the Radboud Data Repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be published after publishing summary data.
Access Criteria: Data will be shared upon reasonable request after signing a data transfer agreement.

REFERENCES:
- [Background] Nieuwhof F, Toni I, Dirkx MF, Gallea C, Vidailhet M, Buijink AWG, van Rootselaar AF, van de Warrenburg BPC, Helmich RC. Cerebello-thalamic activity drives an abnormal motor network into dystonic tremor. Neuroimage Clin. 2022;33:102919. doi: 10.1016/j.nicl.2021.102919. Epub 2021 Dec 16. PMID 34929584
- [Background] Panyakaew P, Cho HJ, Lee SW, Wu T, Hallett M. The Pathophysiology of Dystonic Tremors and Comparison With Essential Tremor. J Neurosci. 2020 Nov 25;40(48):9317-9326. doi: 10.1523/JNEUROSCI.1181-20.2020. Epub 2020 Oct 23. PMID 33097635